CLINICAL TRIAL: NCT04897451
Title: Quality of Life 3 Months After Cervical Ripening
Brief Title: Quality of Life After Cervical Ripening
Acronym: MATUCOL-QOL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Other Study IDs: CHD21-0028
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2021-12

CONDITIONS: Delivery
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with cervical ripening in the context of artificial labor induction
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — EQ5D-5L questionnaire self-reported 3 months after delivery

SUMMARY:
Women's experience of childbirth differs with type of labor, mode of delivery and parity. Induction of labor (IOL) is associated with lower satisfaction of women than spontaneous labor.

A Nigerian study of 252 women with induced labor, irrespective of parity and device used for IOL and a French cohort study of 3042 women with IOL have been published. Theses latter identified several determinants of maternal dissatisfaction.

However, no published study has reported the assessment of quality of life of women at long term after cervical ripening according to the device required for cervical ripening.

The aim of this study is to characterize the quality of life of women after cervical ripening according to parity and device required, and to assess possible factors associated with this quality of life at long-term after delivery.

ELIGIBILITY:
Inclusion Criteria:

- Woman who experienced at least one method of cervical ripening in our hospital

Exclusion Criteria:

- Patient's refusal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Women who experienced at least one method of cervical ripening in our hospital.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
EuroQol 5 Dimension Score | 3 months after delivery
  Quality of life from the EuroQol 5 Dimension questionnaire For each of the dimensions, there are 5 levels coded from 1 to 5. A one-digit number is obtained for each dimension. By combining the 5 dimensions, a 5-digit number is obtained, ranging from 11111 to 55555, representing the health status of the respondent. The code 11111 indicates a person with no problems on the 5 dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume DUCARME, Principal Investigator — CHD Vendee
Locations (1):
- CHD Vendée, La Roche-sur-Yon, France

IPD SHARING:
Plan to Share IPD: No